CLINICAL TRIAL: NCT06136208
Title: Pharmacokinetic Aspects of 25-mg Estradiol Pellet in Climacteric Women Comprehensive Longitudinal Assessment of Release With Estradiol Pellet Analysis (CLARA Study)
Brief Title: Pharmacokinetic Aspects of 25-mg Estradiol Pellet in Climacteric Women
Acronym: CLARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science Valley Research Institute (Other)
Collaborators: Biòs Farmacêutica (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLARA Study
Record Dates: First submitted 2023-10-31; First posted 2023-11-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Climacteric Syndrome; Menopause; Hypoestrogenism
Keywords: Climateric; Estradiol Pellet; Menopause; Pharmacokinectic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: s.c 25 mg estradiol pellet — Subcutaneous insertion of 25 mg estradiol pellet.

SUMMARY:
A single center, prospective, open-label clinical study will be conducted, to monitor serum concentration and pharmacokinetic profile after subcutaneous implantation of a 25mg-estradiol bioabsorbable implant in postmenopausal women.

DETAILED DESCRIPTION:
Assessing serum total estradiol concentration and determination of pharmacokinetic parameters will be performed in participants eligible for the study before and after the insertion of estradiol pellet (25 mg) at different collection times [in the first 24 hours, weekly in the first month and monthly until 6 months are complete]. Additionally, the concentration of other hormones influenced by the action of estradiol will be determined (total testosterone, estrone, FSH, LH, SHBG, and prolactin). Medical visits will be carried out for clinical evaluation and follow-up of the participants in the baseline and after 1 month, 3 months, and 6 months. Assessment of the primary outcome will be performed 6 months after estradiol pellet insertion. N=20 participants.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Woman aged ≥ 41 and ≤ 59 years
* Weight ≥ 50 kg and ≤ 98 kg
* BMI ≥ 18.5 and ≤ 34.9 kg/m²
* Hysterectomy (with or without oophorectomy)
* Serum total estradiol concentration ≤ 50 pg/mL and serum FSH concentration ≥ 25 mIU/mL, both determined by immunoassays
* Presence of menopause-associated symptoms
* Absence of signs and symptoms and propedeutics suggestive of breast cancer evidenced by mammography report (woman aged > 40 years) for less than 12 months = BI-RADS1 or BI-RADS2
* Agreement not to use other hormones (estrogens, androgens and/or progestogens) in any pharmaceutical form during the study

Exclusion Criteria:

* Contraindications to the use of menopausal hormone therapy: Bleeding vaginal of unknown cause; personal history of hormone-dependent neoplasm including breast cancer, precursor lesions of breast cancer; liver disease; porphyria; personal history of coronary artery disease, cerebrovascular and venous thromboembolism; systemic lupus erythematosus with high thromboembolic risk and meningioma
* Comorbidities associated with increased cardiovascular risk: smoking, uncontrolled diabetes, dyslipidemia, and uncontrolled hypertension
* Serious chronic disorders, including metastatic malignancies, kidney disease in the end-stage with or without dialysis, clinically unstable heart disease, or any another disorder that, in the opinion of the investigator, excludes the participant from the study
* Immunocompromise or suspected or confirmed diagnosis of immunodeficiency based on history and/or physical or laboratory examination
* Active liver disease or dysfunction
* Benign or malignant tumors of the liver
* Clinical diagnosis of polycystic ovary syndrome
* Use of other hormones (estrogens, androgens and/or progestogens) in any pharmaceutical form in the last month
* Current use of drugs that alter cytochrome P450 and metabolization of Estrogens
* Current use of tamoxifen, aromatase inhibitors, or agonists/antagonists GnRH for cancer or any other condition
* Current use of phytoestrogens
* Participation in another clinical study within 30 days prior to the start of the Study treatment

Ages: 41 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Serum total estradiol concentration | 0, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days , 21 days , 28 days , 56 days, 84 days, 112 days, 140 days and 168 days
  Multiple blood sample will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days , 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and will be determined by liquid chromatography (LC-MS/MS)
Area under the curve (AUC(0 ∞)) | 0, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days
  Multiple blood sample will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days , 21 days, 28 days, 56 days, 84 days ,112 days ,140 days and 168 days and will be determined by liquid chromatography (LC-MS/MS)
Maximum concentration (Cmax) | 0, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days
  Multiple blood sample will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and will be determined by liquid chromatography (LC-MS/MS)
Time to reach maximum concentration (tmax) | 0, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days
  Multiple blood sample will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and will be determined by liquid chromatography (LC-MS/MS)
Half Life (t1/2) | 0, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days
  Multiple blood sample will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 dyas, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and will be determined by liquid chromatography (LC-MS/MS).

SECONDARY OUTCOMES:
Total testosterone concentration | Pre-insertion of the estradiol pellet; 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days,140 days and 168 days
  Multiple blood will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and total testosterone concentrations will be determined by Liquid chromatography - mass spectrometry
Estrone concentration | Pre-insertion of the estradiol pellet; 2h, 4h, 6h, 8h, 10h, 12, 24h; 7, 14, 21, 28, 56, 84, 112, 140 and 168 days
  Multiple blood will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours , 24 hours; 7 days, 14 days , 21 days , 28days , 56 days, 84 days, 112 days , 140 days and 168 days and estrone concentrations will be determined by LC-MS/MS.
Follicle - stimulating hormone FSH concentration | Pre-insertion of the estradiol pellet; 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days
  Multiple blood will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and Follicle-stimulating hormone concentrations will be determined by electrochemiluminescence
Luteinizing hormone - hormone LH concentration | Pre-insertion of the estradiol pellet; 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days
  Multiple blood will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and Follicle-stimulating hormone concentrations will be determined by electrochemiluminescence
Sex hormone binding globulin SHBG concentration | Pre-insertion of the estradiol pellet; 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days
  Multiple blood will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days,28 dyas, 56 days, 84 days, 112 days, 140 days and 168 days and Follicle-stimulating hormone concentrations will be determined by electrochemiluminescence
Prolactin concentration | Pre-insertion of the estradiol pellet; 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days
  Multiple blood will be collected before pellet implantation and 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 7 days, 14 days, 21 days, 28 days, 56 days, 84 days, 112 days, 140 days and 168 days and Follicle-stimulating hormone concentrations will be determined by electrochemiluminescence

OTHER OUTCOMES:
Adverse events | pre-insertion of the estradiol pellet; 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours; 28 days, 84 days, and 168 days
  Number of participants experiencing serious adverse events (SAEs) and adverse events leading to discontinuation in the study. Adverse events reported by study participants (any including non-serious ones)
Change from baseline in the Menopause Rating Scale (MRS) score (global, psychological, somatic, and urogenital domains evaluated in clinical visits | 28 days, 84 days, and 168 days post-insertion of the estradiol pellet
  The MRS is a patient reported assessment of 11 symptoms of menopause on a scale of 0 (none) to 4 (very severe). The MRS groups symptoms into three subscales: psychological, somatic, and urogenital. A composite score is calculated by adding the items in each dimension (subscale). The total score is the sum of the three dimensional scores. A higher score indiactes a greater severity of perceived menopausal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: André Luiz Malavasi de Oliveira Longo, MD, PhD, Study Chair — Science Valley Research Institute
Locations (1):
- Irmandade Da Santa Casa De Misericórdia De Santos - Science Valley Research Center, Santos, São Paulo, Brazil

REFERENCES:
- [Background] Casals G, Costa RF, Rull EU, Escobar-Morreale HF, Argente J, Sesmilo G, Biagetti B. Recommendations for the measurement of sexual steroids in clinical practice. A position statement of SEQCML/SEEN/SEEP. Adv Lab Med. 2023 Mar 9;4(1):52-69. doi: 10.1515/almed-2023-0020. eCollection 2023 Apr. PMID 37359897
- [Background] del Carmen Cravioto M, Larrea F, Delgado NE, Escobar AR, Diaz-Sanchez V, Dominguez J, de Leon RP. Pharmacokinetics and pharmacodynamics of 25-mg estradiol implants in postmenopausal Mexican women. Menopause. 2001 Sep-Oct;8(5):353-60. doi: 10.1097/00042192-200109000-00010. PMID 11528362
- [Background] Hamoda H, Panay N, Pedder H, Arya R, Savvas M. The British Menopause Society & Women's Health Concern 2020 recommendations on hormone replacement therapy in menopausal women. Post Reprod Health. 2020 Dec;26(4):181-209. doi: 10.1177/2053369120957514. Epub 2020 Oct 12. No abstract available. PMID 33045914
- [Background] Kuhl H. Pharmacology of estrogens and progestogens: influence of different routes of administration. Climacteric. 2005 Aug;8 Suppl 1:3-63. doi: 10.1080/13697130500148875. PMID 16112947
- [Background] Lobo RA, March CM, Goebelsmann U, Krauss RM, Mishell DR Jr. Subdermal estradiol pellets following hysterectomy and oophorectomy. Effect upon serum estrone, estradiol, luteinizing hormone, follicle-stimulating hormone, corticosteroid binding globulin-binding capacity, testosterone-estradiol binding globulin-binding capacity, lipids, and hot flushes. Am J Obstet Gynecol. 1980 Nov 15;138(6):714-9. PMID 6776814
- [Background] Lobo RA. Hormone-replacement therapy: current thinking. Nat Rev Endocrinol. 2017 Apr;13(4):220-231. doi: 10.1038/nrendo.2016.164. Epub 2016 Oct 7. PMID 27716751
- [Background] Manson JE, Bassuk SS, Kaunitz AM, Pinkerton JV. The Women's Health Initiative trials of menopausal hormone therapy: lessons learned. Menopause. 2020 Aug;27(8):918-928. doi: 10.1097/GME.0000000000001553. PMID 32345788
- [Background] Notelovitz M, Johnston M, Smith S, Kitchens C. Metabolic and hormonal effects of 25-mg and 50-mg 17 beta-estradiol implants in surgically menopausal women. Obstet Gynecol. 1987 Nov;70(5):749-54. PMID 3658285
- [Background] Owen EJ, Siddle NC, McGarrigle HT, Pugh MA. 25 mg oestradiol implants--the dosage of first choice for subcutaneous oestrogen replacement therapy? Br J Obstet Gynaecol. 1992 Aug;99(8):671-5. doi: 10.1111/j.1471-0528.1992.tb13853.x. PMID 1327094
- [Background] Stanczyk FZ, Shoupe D, Nunez V, Macias-Gonzales P, Vijod MA, Lobo RA. A randomized comparison of nonoral estradiol delivery in postmenopausal women. Am J Obstet Gynecol. 1988 Dec;159(6):1540-6. doi: 10.1016/0002-9378(88)90591-1. PMID 3144919
- [Background] Stuenkel CA, Davis SR, Gompel A, Lumsden MA, Murad MH, Pinkerton JV, Santen RJ. Treatment of Symptoms of the Menopause: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2015 Nov;100(11):3975-4011. doi: 10.1210/jc.2015-2236. Epub 2015 Oct 7. PMID 26444994
- [Background] Suhonen SP, Allonen HO, Lahteenmaki P. Sustained-release subdermal estradiol implants: a new alternative in estrogen replacement therapy. Am J Obstet Gynecol. 1993 Nov;169(5):1248-54. doi: 10.1016/0002-9378(93)90291-p. PMID 8238193
- [Background] Thom MH, Collins WP, Studd JW. Hormonal profiles in postmenopausal women after therapy with subcutaneous implants. Br J Obstet Gynaecol. 1981 Apr;88(4):426-33. doi: 10.1111/j.1471-0528.1981.tb01008.x. PMID 6784745